CLINICAL TRIAL: NCT01537770
Title: Percutaneous Vertebroplasty Opposite - Infiltration of the Periost and Vertebral Body With Lidocaine - as Pain Palliative Treatment of Osteoporotic Vertebral Fractures of the Thoracic and Lumbar Spine
Brief Title: Vertebroplasty Compared With a Sham-procedure for Painful Acute Osteoporotic Vertebral Fractures
Acronym: VOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Emil Jesper Hansen, MD, PhD, Spine Centre of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-024050-10
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Osteoporotic Fractures
Keywords: Vertebroplasty; Low energy osteoporotic vertebral fractures; of the thoracic and/or lumbar spine
MeSH Terms: conditions — Osteoporotic Fractures | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vertebroplasty (Active Comparator): Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. Bone cement is prepared on the bench and injected under constant fluoroscopy into the vertebral body. Injection is stopped when the cement reaches to the posterior aspect of the vertebral body or leaks into an extraosseous space, such as the intervertebral disk or an epidural or paravertebral vein.
  Interventions: Procedure: Percutaneous vertebroplasty
- lidocaine injection (Sham Comparator): Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. 2 ml of 1% Lidocaine is injected in each needle. Bone cement is prepared on the bench simulating the vertebroplasty-procedure.
  Interventions: Procedure: Lidocaine injection

INTERVENTIONS:
Procedure: Percutaneous vertebroplasty — Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. Bone cement is prepared on the bench and injected under constant fluoroscopy into the vertebral body. Injection is stopped when the PMMA reaches to the posterior aspect of the vertebral body or leaks into an extraosseous space, such as the intervertebral disk or an epidural or paravertebral vein.
  Arms: Vertebroplasty
Procedure: Lidocaine injection — Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. 2 ml of 1% Lidocaine is injected in each needle. Bone cement is prepared on the bench simulating the vertebroplasty-procedure.
  Arms: lidocaine injection

SUMMARY:
The main purpose of this study:

- to determine whether vertebroplasty has a pain palliating effect superior to a sham-procedure for acute painful osteoporotic vertebral fractures of the thoracic and lumbar spine.

Secondary purposes:

* To determine if there are differences in the two methods on preventing forward tilting of the spine and/or shortening of the total height of the spine.
* measure if there are differences in change of lung capacity between the two methods

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy of bone cement injection (PVP) for patients with acute painful osteoporotic compression fractures, as compared with a simulated procedure with injection of Lidocaine. Our hypothesis is, that patients who had undergone PVP would report less pain during the first 1-12 weeks and at 12 months (primary outcomes) than those in the sham control group.

The study design of VOPE is a single center double blinded RCT concerning the treatment of patients with a painful osteoporotic VCF. Patients are referred to the principal investigator at Middelfart hospital from the emergency rooms, orthopedics departments, GP's and chiropractors from the Region of Southern Denmark. Prior to enrolling patients randomization-envelopes are constructed in blocks of 20. Upon obtaining informed consent, a study-number is assigned to each patient. The final randomization for each patient, takes place in the operation room upon opening the sealed envelope deciding which of the two operations are to be performed. A total of 80 patients will be enrolled, 40 in each group. This is based on the assumption of a 2.0 point difference in pain relief (VAS Score) and a maximum of 35% withdrawal rate (α=0.05 and β=0.20). The enrolment of patients will take place in a single center, the spine surgery department of Middelfart hospital in Denmark. Randomization will start February 2012 with an expected completion of enrolment by May 2013. There is a one-year follow-up, with the possibility of an extended follow-up at two years.

The overall Institutional Review Board approval is obtained at Middelfart Hospital.

Osteoporosis- and pain medication:

All patients are, in cooperation with the osteoporosis clinic at Odense University Hospital (OUH), DXA-scanned 3 times during the follow-up period, and receives, regarding these results, the correct antiosteoporotic treatment determined by a endocrinology senior consultant. Analgesics are classified following the WHO classification: (1) Paracetamol (acetaminophen), (2) Tramadol, (3) Tramadol and Paracetamol, (4) Morphine.

Clinical follow-up:

An experienced nurse-practitioner and research consultant requests patients to fill out a standard questionnaire before and at 1 day, 1-11 weeks, and 3 and 12 months after the procedure. The patients will receive a folder including questionnaires for each of the first 11 weeks and will be contacted by telephone once every week and asked to fill out the questionnaires. The questionnaire consist of the VAS and NRS score and questions about use of pain medication. The VAS score is a 10 cm line pain score ranging from "no pain" to "worst pain ever", the NRS is a similar tool where patients are asked in 3 different ways to describe their pain between 0 and 10 where 10 is the worst pain ever. Other medical treatment is registered at 0, 3 and 12 months.

Secondary outcomes are back pain related disability and QOL as measured with the SF-36 Questionnaire and the EuroQol 5D Questionnaire. The EQ5D score ranges from 0 (worst quality of life) to 1 (best quality of life). This questionnaire will be completed at three measurement moments (before and at 3, and 12 months after the procedure). SF-36 scores from 0-100, (100 as the best outcome), 4 domains describing tghe physical function and 4 describing mental health. The lung capacity will be measured by the principal investigator with a spirometer at before and at 3 and 12 months.

Statistical analysis:

The data will be analysed according to the intention-to-treat principle. Standard statistical techniques will be used to describe characteristics of patients in both groups using the STATA programme. If incomparability appears at baseline, we will in secondary analysis adjust for differences. The primary outcome, significant pain relief will be compared with the analysis of variance for repeated measures. If adjustment for possible baseline incomparability is needed, analysis of covariance will be done.

ELIGIBILITY:
Inclusion Criteria:

* VCF on X-ray of the spine (minimal 15% loss of height) level of VCF Th6 or lower
* back pain ≤ 8 weeks at time of surgery
* ≥ 50 years of age
* bone edema on MRI of the fractured vertebral body
* focal tenderness on VCF level

Exclusion Criteria:

* severe cardio-pulmonary condition
* untreatable coagulopathy
* systemic or local infection of the spine (osteomyelitis, spondylodiscitis)
* suspected alternative underlying disease (malignancy)
* radicular and/or cauda compression syndrome
* contra-indication for MRI

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pain relief | 12 Months
  Primary outcome will be pain relief at 1 day, 1-12 weeks, and 12 months. The questionnaire consist of the VAS score and questions about use, ammount and type of pain medication. Patients are asked to fill out the VAS and NRS score, and use of analgesics is recorded once every week during the first 3 months after randomization.

SECONDARY OUTCOMES:
Quality of life EQ5D | 12 months
  Quality of life as meassured with the EuroQol 5D questionnaire at 3 and 12 months. It consists of 5 different questions.
Physical function, disability etc. | 12 months
  The patients fill out the SF-36 questionnaire at baseline and at 3 and 12 months. It consists of 36 questions containing 8 domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning,emotional role functioning, social role functioning, mental health.
Lung capacity | 12 months
  Lungcapacity as examined with a spirometer at 3 and 12 months. The patients history of lungdiseases and use of medicin affecting the lungcapacity is registered at baseline and at 3 and 12 months.
Subsidence of the affected vertebral bodies and local kyphosis | 12
  X-ray images of the entire spine, lateral view at 3 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Ø Andersen, MD, associate Professor, Study Chair — Sygehus Lillebaelt; Emil J Hansen, MD, PhD student, Principal Investigator — Sygehus Lillebaelt; Rikke Rousing, PhD, Study Director — Sygehus Lillebaelt; Hans Tropp, MD, Professor, Study Chair
Locations (1):
- Middelfart Spinesurgery research department, Middelfart, Region Syddanmark, Denmark